CLINICAL TRIAL: NCT06128876
Title: Artificial Intelligence-based Risk Stratification and Mid-term Outcomes in Severe Aortic Stenosis: Insights from Cardiac Magnetic Resonance Imaging
Brief Title: CMR-AI and Outcomes in AS
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Matthias Koschutnik, Principal Investigator, Medical University of Vienna
Other Study IDs: VIE_CMR-AI
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis; Artificial Intelligence; Cardiac Magnetic Resonance; Imaging; Outcomes
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background & Aims: Artificial Intelligence (AI) in cardiac magnetic resonance (CMR) imaging has previously been shown to provide highly reproducible and accurate measures of myocardial structure and function, outperforming clinical experts. The prognostic value of more sensitive markers of early left (LV) and right ventricular (RV) function, such as global longitudinal shortening (GLS), mitral annular plane systolic excursion (MAPSE), and tricuspid annular plane systolic excursion (TAPSE) has not been established due to the lack of automated analysis. Thus, our aim is to evaluate whether AI-based measurements of these early markers of adverse cardiac remodeling convey relevant prognostic information in patients with severe aortic stenosis (AS) beyond LV and RV ejection fraction (EF).

Materials & Methods: In a current large-scale international, prospective, multi-center study ~1500 patients with severe AS underwent CMR imaging prior to aortic valve replacement (AVR). An AI-based algorithm, developed in the UK, was used for fully automated assessment of parameters of cardiac structure (end-diastolic volume, end-systolic volume, LV mass, maximum wall thickness) and function (EF, GLS, MAPSE, TAPSE). In this proposed follow-up project, we aim to associate these AI-based CMR parameters at baseline with mid-term clinical outcomes at 24-months post-AVR. A composite of all-cause mortality and heart failure hospitalization will serve as the primary endpoint. CMR-AI will be repeated at 24-months follow-up and trajectories from pre- to post-AVR will be assessed as a secondary endpoint.

Future Outlook: In severe AS, a novel AI-based algorithm allows immediate and precise measurements of ventricular structure and function on CMR imaging. Our goal is to identify early markers of cardiac dysfunction indicating adverse mid-term prognosis post-AVR. This has guideline-forming potential as the optimal timepoint for AVR in patients with AS is currently a matter of debate.

DETAILED DESCRIPTION:
Artificial Intelligence (AI) and Machine Learning are reshaping our daily clinical practice, which has the potential to be more efficient, precise, and personalized. Adopting these technologies in cardiac imaging does not only affect decision making by improved accuracy and risk stratification but also significantly reduces scan times and post-imaging workup.

Current guidelines acknowledge cardiac magnetic resonance (CMR) imaging as gold standard for assessment of myocardial structure and function. Despite the fundamental importance in various cardiac diseases, measurements of size, mass, and ejection fraction (EF) are flawed by the inherent variability and subjectivity of human analysis. Recent developments in deep learning using convolutional neural networks (CNNs) allow for automated segmentation of the ventricular blood pool and myocardium using pre-existing CMR datasets. Importantly, these tools are integrated into CMR scanners generating real-time measurements without the need of time-consuming image post-processing. AI-based models have previously shown similar to superior precision in ventricular contouring, volumetry, and maximum wall thickness (MWT) measurements, outperforming clinical experts.

In patients with aortic stenosis (AS), changes in EF more often occur late in the disease process, whereas longitudinal shortening represents an earlier and more sensitive marker of left ventricular (LV) dysfunction. However, these CMR measurements are subjective, time-consuming, and therefore not routinely performed due to the lack of automated analysis. Recently, AI-measured global longitudinal shortening (GLS) and mitral annular plane systolic excursion (MAPSE) have been demonstrated to provide more reproducible and accurate results compared to human experts. We hypothesize that AI-based GLS and MAPSE could convey important prognostic information beyond LVEF in severe AS and represent early markers of adverse cardiac remodeling and outcome following aortic valve replacement (AVR). Furthermore, in our own working group, we could demonstrate that right ventricular (RV) dysfunction on CMR, rather than conventional parameters assessed by echocardiography, was independently associated with outcome in individuals with AS undergoing transcatheter aortic valve implantation. We aim to extend on our findings and investigate whether AI-based RV GLS and tricuspid annular plane systolic excursion (TAPSE) represent early markers of RV dysfunction indicating adverse prognosis.

Finally, the assessment of reverse cardiac remodeling by CMR requires reproducibility. AI has been proven to outperform humans in both precision and accuracy, and therefore has great potential for the comprehensive evaluation of longitudinal structural changes in AS following AVR. We aim to analyze mid-term reverse cardiac remodeling in patients with AS using novel AI technology.

Aims

With significant previous contributions in cardiac imaging and valvular heart disease being made by our research group, we aim to provide automated, precise, and time-saving algorithms to identify patients at risk post-AVR by addressing the following:

* Association of AI-measured LV and RV structural and functional markers on CMR prior to AVR with mid-term clinical outcomes at 24-months following AVR.
* Reverse cardiac remodeling, as determined by CMR-AI parameters, at baseline versus 24-months after AVR.

Methods

This project is designed as a large-scale international, prospective, multi-center, longitudinal-observational cohort study aimed at identifying predictors of structural and functional recovery in patients with severe AS undergoing clinically indicated AVR. Participants were previously enrolled from seven university-affiliated tertiary care centers in Continental Europe, the UK, and Asia between January 2020 and August 2024.

Baseline evaluation consisted of comprehensive pre-operative cardiac phenotyping including quality of life assessment, blood tests, electrocardiogram (ECG), and imaging (CMR and echocardiography). For this proposed project, reverse cardiac remodeling and mid-term clinical outcomes will be evaluated 24-months post-AVR through repeat baseline investigations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Severe AS scheduled for Heart Team decision

Exclusion Criteria:

* Inability or unwillingness to perform any of the diagnostic tests
* Inability or unwillingness to participate in follow-up visits
* Metal implants, e.g. cochlear implants and pacemakers
* Chronic kidney failure (GFR < 30 ml/min/1.73m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe degenerative AS scheduled for valvular treatment undergoing pre-procedural CMR imaging were previously enrolled from seven university-affiliated tertiary care centers in Continental Europe, the UK, and Asia between January 2020 and August 2024.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with AI-measured parameters of impaired left and right ventricular structure and function on cardiac magnetic resonance imaging and association with the composite of all-cause death and heart failure hospitalization. | 2 years
  Association of AI-based parameters (end-diastolic volume [ml], end-systolic volume [ml], left ventricular mass [gram], maximum wall thickness [mm], ejection fraction [%], global longitudinal shortening [%], mitral/tricuspid annular plane systolic excursion [mm]) on cardiac magnetic resonance imaging with the composite of all-cause death and heart failure hospitalization.
  Captured clinical endpoints will include all-cause death, cardiovascular mortality, and heart failure hospitalization. Data will be ascertained by follow-up visits, state-wide electronic hospital charts, and phone calls. In addition, mortality data will be obtained via National Death Registries of the participating countries.

SECONDARY OUTCOMES:
Number of patients with AI-measured parameters of impaired left and right ventricular structure and function on cardiac magnetic resonance imaging and association with components of the primary endpoint analyzed individually. | 2 years
  Association of AI-based parameters (end-diastolic volume [ml], end-systolic volume [ml], left ventricular mass [gram], maximum wall thickness [mm], ejection fraction [%], global longitudinal shortening [%], mitral/tricuspid annular plane systolic excursion [mm]) on cardiac magnetic resonance imaging with components of the primary endpoint (all-cause death and heart failure hospitalization) analyzed individually.
  Captured clinical endpoints will include all-cause death, cardiovascular mortality, and heart failure hospitalization. Data will be ascertained by follow-up visits, state-wide electronic hospital charts, and phone calls. In addition, mortality data will be obtained via National Death Registries of the participating countries.
Number of patients with AI-measured parameters of impaired left and right ventricular structure and function on cardiac magnetic resonance imaging and association with cardiovascular mortality. | 2 years
  Association of AI-based parameters (end-diastolic volume [ml], end-systolic volume [ml], left ventricular mass [gram], maximum wall thickness [mm], ejection fraction [%], global longitudinal shortening [%], mitral/tricuspid annular plane systolic excursion [mm]) on cardiac magnetic resonance imaging with cardiovascular mortality.
  Captured clinical endpoints will include all-cause death, cardiovascular mortality, and heart failure hospitalization. Data will be ascertained by follow-up visits, state-wide electronic hospital charts, and phone calls. In addition, mortality data will be obtained via National Death Registries of the participating countries.

OTHER OUTCOMES:
Number of patients with AI-measured parameters of impaired left and right ventricular structure and function on cardiac magnetic resonance imaging at baseline and changes at 2-year follow-up after aortic valve replacement (AVR). | 2 years
  Longitudinal trajectories of AI-based parameters (end-diastolic volume [ml], end-systolic volume [ml], left ventricular mass [gram], maximum wall thickness [mm], ejection fraction [%], global longitudinal shortening [%], mitral/tricuspid annular plane systolic excursion [mm]) on cardiac magnetic resonance imaging from pre- to 2-year post-AVR.
  Captured clinical endpoints will include all-cause death, cardiovascular mortality, and heart failure hospitalization. Data will be ascertained by follow-up visits, state-wide electronic hospital charts, and phone calls. In addition, mortality data will be obtained via National Death Registries of the participating countries. CMR will be repeated at 2 year.

CONTACTS AND LOCATIONS:
Locations (7):
- Medical University of Vienna, Vienna, Austria
- Université Catholique de Louvain, Brussels, Belgium
- University of Goettingen Medical Center, Göttingen, Germany
- Vilnius University, Vilnius, Lithuania
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University College, Seoul
- Barts Heart Centre, London, United Kingdom